CLINICAL TRIAL: NCT07115953
Title: Sub-study of SPYRAL AFFIRM: Streamlined Denervation With spYral For an Optimized Treatment (SPYRAL SWYFT)
Brief Title: Streamlined Denervation With spYral For an Optimized Treatment (SPYRAL SWYFT) in Subjects With Uncontrolled Hypertension
Acronym: SWYFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT20044RDN004_SWYFT; SPYRAL AFFIRM (NCT05198674) (Other: ClinicalTrials.gov); CIV-21-09-037767 (Other: EUDAMED)
Record Dates: First submitted 2025-07-24; First posted 2025-08-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases; Chronic Kidney Diseases; Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases; Renal Insufficiency, Chronic; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SWYFT cohort (Experimental): Renal angiography and Renal Denervation (Symplicity Spyral™ multi-electrode renal denervation system)
  Interventions: Device: Symplicity Spyral™ multi-electrode renal denervation system

INTERVENTIONS:
Device: Symplicity Spyral™ multi-electrode renal denervation system — After a renal angiography according to standard procedures, subjects are treated with the renal denervation procedure.
  Other Names: Renal Angiography; Renal Denervation

SUMMARY:
The purpose of the SPYRAL SWYFT sub-study is to evaluate whether renal denervation with the Symplicity Spyral system performed in the main and first order branch renal arteries yields a shorter procedure time and is as effective in reducing blood pressure than the procedural approach used in the SPYRAL HTN-ON MED and SPYRAL PIVOTAL - SPYRAL HTN-OFF MED clinical studies in an uncontrolled hypertensive population.

DETAILED DESCRIPTION:
SPYRAL SWYFT will evaluate the long-term safety, efficacy, and durability of the Symplicity Spyral system to determine whether renal denervation performed in the main and first order branch renal arteries yields a shorter procedure time and is as effective in reducing blood pressure than the procedural approach used in the SPYRAL HTN-ON MED and SPYRAL PIVOTAL - SPYRAL HTN-OFF MED clinical studies (where all accessible renal arterial vessels between 3 and 8 mm in diameter including accessory, branch and main renal arteries (outside the kidney parenchyma) were targeted for ablation).

SPYRAL SWYFT study is conducted under the overarching SPYRAL AFFIRM protocol (NCT05198674), focused on EU and APAC regions.

ELIGIBILITY:
Inclusion Criteria:

1. Individual is diagnosed with hypertension and has a baseline office systolic blood pressure ≥140 mmHg
2. Individual has a baseline office diastolic blood pressure ≥ 90 mmHg
3. Individual has an average systolic baseline home blood pressure ≥135 mmHg (with ≥7 days of valid pre-procedure measurements)
4. Individual has a valid 24-hour Ambulatory Blood Pressure Measurement at baseline

Exclusion Criteria:

1. Individual lacks appropriate renal artery anatomy
2. Individual has undergone prior renal denervation
3. Individual has a documented condition that would prohibit or interfere with ability to obtain an accurate blood pressure measurement
4. Individual requires chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea
5. Individual has an estimated glomerular filtration rate (eGFR) of <45 mL/min/1.73m2
6. Individual has one or more episode(s) of orthostatic hypotension
7. Individual is pregnant, nursing or planning to become pregnant
8. Individual has documented primary pulmonary hypertension
9. Individual has documented type 1 diabetes mellitus or poorly-controlled type 2 diabetes mellitus with glycosylated hemoglobin greater than 8.0%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Procedure time | Procedure
  Procedure time will be compared to the SPYRAL HTN-ON MED and SPYRAL PIVOTAL - SPYRAL HTN-OFF MED procedure times.
Office Systolic Blood Pressure Change | 6 months
  Office Systolic Blood Pressure (OSBP) change from baseline to 6 months will be compared to the SPYRAL HTN-ON MED and SPYRAL PIVOTAL - SPYRAL HTN-OFF MED study efficacy endpoints using a propensity score stratified baseline blood pressure adjusted analysis at 3 months (OFF MED) and 6 months (ON MED).

SECONDARY OUTCOMES:
Office Systolic Blood Pressure change | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Home Blood Pressure change | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Change in blood pressure as measured by 24-hour ABPM | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Percent of subjects achieving blood pressure control as measured by OBP, HBP and ABPM | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Time subject's blood pressure is controlled | Procedure to 36 months post-procedure
Change in number of anti-hypertensive medications taken from baseline | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Change from baseline in hypertension health status score | From baseline to 3, 6, 12, 24, and 36 months post-procedure. A higher score means a better outcome.
Evaluate factors influencing blood pressure response to renal denervation | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Evaluation of slope of eGFR | From baseline to 3, 6, 12, 24, and 36 months post-procedure
Incidence of safety events, including major adverse events | From baseline to 3, 6, 12, 24, and 36 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: David Lee, MD, Principal Investigator — Stanford University; Konstantinos Tsioufis, Prof Dr, Principal Investigator — Hippokration General Hospital of Athens
Locations (16):
- Australia (2):
  - The Alfred Hospital, Melbourne
  - Royal Perth Hospital, Perth
- Belgium (5):
  - Ziekenhuis Oost Limburg - Campus Sint-Jan, Genk, Limburg
  - CHC MontLégia, Liège, Liège
  - Algemeen Stedelijk Ziekenhuis - Campus Aalst, Aalst
  - AZ Sint Jan Brugge-Oostende av, Bruges
  - Universitair Ziekenhuis Gent, Ghent
- Germany (4):
  - Universitat des Saarlandes, Homburg, Saarland
  - Sana Kliniken Lübeck GmbH, Lübeck, Schleswig-Holstein
  - Universitätsklinikum Erlangen, Erlangen
  - Leipzig Heart Institute, Leipzig
- Mater Misericordiae University Hospital, Dublin, Dublin, Ireland
- Netherlands (2):
  - Zuyderland Medisch Centrum Heerlen, Heerlen
  - Erasmus University Medical Center, Rotterdam
- National Taiwan University Hospital, Taipei, Taiwan
- Oxford University Hospitals NHS Trust - John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data. Aggregate results will be made publicly available via publications and conference presentations.